CLINICAL TRIAL: NCT03434171
Title: Effect of Aerobic Exercises With Selected Phytoestrogen Product on Hot Flushes in Post-menopausal Women
Brief Title: Effect of Aerobic Exercises With Selected Phytoestrogens on Hot Flushes in Menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Intervention Model Description: What is the effect of aerobic exercises with diet modification on hot flushes, lutenizing hormone (L.H) and follicle stimulating hormone (F.S.H) in post-menopausal women
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic excercise (Active Comparator): women who practiced treadmill exercise program for 30 minutes at 60% to 70% of maximum heart rate. The treatment sessions will be repeated 3 times per week for 12 weeks
  Interventions: Behavioral: Aerobic excercise; Dietary Supplement: soy products
- Dietary modfications (Active Comparator): women who received diet modification contains soy products (phytoestrogen) such as soy milk and soy beans every day for 12 weeks only
  Interventions: Dietary Supplement: soy products

INTERVENTIONS:
Behavioral: Aerobic excercise — practiced treadmill exercise program for 30 minutes at 60% to 70% of maximum heart rate. The treatment sessions will be repeated 3 times per week for 12 weeks
  Other Names: trademill
  Arms: Aerobic excercise
Dietary Supplement: soy products — diet modification contains soy products (phytoestrogen) such as soy milk and soy beans every day for 12 weeks only

SUMMARY:
50 menopausal women with the diagnosis of hot flushes were randomized to 1 of 2 groups

Group (A):

It consists of 25 women who practiced treadmill exercise program for 30 minutes at 60% to 70% of maximum heart rate. The treatment sessions will be repeated 3 times per week for 12 weeks.

Group (B):

It consists of 25 women who received diet modification contains soy products (phytoestrogen) such as soy milk and soy beans every day for 12 weeks only.

DETAILED DESCRIPTION:
50 menopausal women with the diagnosis of hot flushes were randomized to 1 of 2 groups

Group (A):

It consists of 25 women who practiced treadmill exercise program for 30 minutes at 60% to 70% of maximum heart rate. The treatment sessions will be repeated 3 times per week for 12 weeks.

Group (B):

It consists of 25 women who received diet modification contains soy products (phytoestrogen) such as soy milk and soy beans every day for 12 weeks only.

ELIGIBILITY:
Inclusion Criteria:

* menopausal women minimum 2 years after menopause Patients were required to have at least moderate hot flashes at time of randomization, having a score ≥ 40 in Hot Flash-Related Daily Interference Scale (HFRDIS)

Exclusion Criteria:

* women with BMI > 30kg/m2 ingestion of any psychotropic and antidepressant medications, any Selective Estrogen Receptor Modulator medications (e.g., tamoxifen and raloxifen), any Aaromatase inhibitor medications (e.g., anastrozole, letrozole, and exemestane), leuprolide acetate, clonidine, gabapentin, pregabalin, amino acid supplements, over the counter (OTC) medications that reduced hot flashes during the last 4 weeks, ingestion of estrogen and progesterone based medications, history of suicidal thoughts, substance or alcohol dependence (with the exception of nicotine dependence) during the last 3 months and Electroconvulsive therapy (ECT) during the last 2 months.

Ages: 47 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Heat sensation changes | 12 weeks after excercise
  the severity of hot flashes score changes

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided